CLINICAL TRIAL: NCT00388908
Title: Addressing Vertebral Osteoporosis Incidentally Detected to Prevent Future Fractures: The AVOID FRACTURE Study
Brief Title: Addressing Vertebral Osteoporosis Incidentally Detected to Prevent Future Fractures
Acronym: AVOID Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIHR-MOP-79325
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2015-07

CONDITIONS: Osteoporosis
Keywords: vertebral fractures; osteoporosis; prevention; case-finding; quality improvement
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Counseling

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Multifaceted intervention
  Interventions: Behavioral: Reminders and opinion leader generated guidelines +/- leaflets and counselling
- B (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Reminders and opinion leader generated guidelines +/- leaflets and counselling
  Arms: A
Other: Usual Care
  Arms: B

SUMMARY:
Osteoporosis is a common and progressive condition that leads to broken bones (fractures), which cause pain, disability, deformity, and even death. There are new treatments available that can decrease the risk of a fracture by 50%, and the people who benefit the most are those with osteoporosis who have already had a fracture, like a vertebral (spine) fracture. Vertebral fractures are usually "silent," and ~20% of people over the age of 60 years have had one although they don't know it. Many of these people have had chest x-rays done for other reasons, and these x-rays can incidentally detect these silent fractures. Although most people with a vertebral fracture should be tested and treated for osteoporosis, studies demonstrate that less than one-quarter of older people with a vertebral fracture are ever investigated or even treated. This reflects a gap between evidence-based best practice and everyday practice in the community. The proposed research addresses this care-gap by using a quality improvement intervention that uses chest x-rays done in the Emergency Department to remind family physicians about osteoporosis while providing them with evidence-based treatment guidelines - with or without educating and empowering patients about osteoporosis. The effectiveness of this intervention will be compared to usual care in a controlled trial. The intent of this research is to improve quality of care for patients at high risk of fracture, by increasing rates of testing and treatment of osteoporosis.

DETAILED DESCRIPTION:
Objective: To improve the quality of care for elderly patients with osteoporosis and vertebral fractures incidentally detected by a chest radiograph in the Emergency Department.

Background: Osteoporosis leads to decreased bone mass, skeletal fragility, and fractures. Osteoporosis affects at least 1.4 million Canadians, 25% of women and 12% of men >60 years of age. The most common osteoporotic fractures are vertebral (spinal), two-thirds of which are asymptomatic. Irrespective of symptoms, these "silent" fractures cause disability, deformity, and death. Compared to those with normal bones and no fracture, the patient with osteoporosis and vertebral fracture has a 20-fold increased risk of future fracture. Guidelines recommend aggressive treatment because rate of re-fracture is 20% within 1 year and treatment reduces risk by 40-50%. Guidelines do not, however, recommend population screening for vertebral fractures. We reported (Arch Intern Med, 2005) that chest radiographs performed in the Emergency Department detected "incidental" fractures in 16% of elderly patients, although only 25% of patients were treated for osteoporosis. The care gap between evidence-based best practice and usual care needs to be urgently addressed.

Hypothesis: The proposed intervention will improve rates of diagnosis and treatment of osteoporosis in high-risk patients. The intervention will be directed at physicians (patient-specific reminders and opinion leader generated 1-page guidelines) with or without patient-activation (leaflets and telephone-based counseling).

Specific Aims: To determine whether exposure to a physician-directed quality improvement intervention can- Aim #1. Increase rates of osteoporosis treatment in patients with newly recognized vertebral fracture(s); Aim #2. Increase patients' self-reported diagnosis of osteoporosis and other related knowledge; Aim #3. Be further augmented by the addition of patient-activation.

Study Design: A single-center prospective nonrandomized controlled trial with blinded (allocation-concealed) ascertainment of outcomes comparing the proposed physician-intervention to usual care controls. We define usual care as notification of the patients' physician of chest radiograph results. Allocation will be on the basis of an alternate-week time series design, with the proposed intervention "on" for all patients for one week, followed by the intervention being "off" (i.e., usual care) the next week. After 3 months, controls will be offered the physician-intervention plus patient-activation, with outcomes recollected 3 months later. Eligible patients will be >60 years of age who present to the Emergency Department: (1) with a chest radiograph reporting the presence of a vertebral fracture, (2) are not taking prescription osteoporosis treatment, and (3) are discharged home. The primary outcome is the proportion of patients starting prescription osteoporosis treatment within 3 months of fracture recognition; secondary outcomes include BMD testing and diagnosis of osteoporosis. The intervention is expected to increase the primary outcome by at least 20% (absolute) over usual care rates of 10%. With alpha=0.05, beta=0.80, 20% losses-to-followup, and additional power to address secondary outcomes and effects of patient-activation, the required sample size is 240 patients.

Pilot Data and Feasibility: Our pilot study (AJR, 2004) found institutional true-positive reporting rates for vertebral fractures were 60%, with 100% specificity, compared with reference standard. A 1-year feasibility study of a random sample of ~5000 radiographs was then undertaken (Arch Intern Med, 2005). Based on these data, we expect to enroll 3-4 patients/week, complete recruitment in ~20 months, ascertain outcomes by 30 months, and finish the study in 3 years. The research team has generated pilot data, systematically reviewed pertinent literature, recruited opinion leaders to create guidelines, trained research staff, refined methods for outcomes ascertainment; and conducted related studies of wrist (Annals Intern Med, 2004) and hip fractures.

Significance: To our knowledge, there are no studies examining strategies to improve care for this vulnerable and high-risk population, and we believe our results will be important regardless of findings. If "negative" it will provide evidence that more costly and laborious interventions will be needed to overcome clinical inertia; if positive, however, our intervention should be widely applicable. In addition, positive results can be easily extended to other related populations (e.g., routine chest radiographs done for admission to nursing homes) and can be adapted for implementation via other modalities (e.g., computerized decision support, telemedicine).

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or greater
* chest radiograph that reports the presence of a vertebral fracture
* discharged home.

Exclusion Criteria:

* unable to provide simple informed consent or unwilling to participate in the study
* unable to read, understand, and converse in English
* admitted to hospital
* currently enrolled in the pilot study or other osteoporosis-related studies
* currently taking any prescription osteoporosis treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the proportion of patients starting prescription osteoporosis treatment within 3 months of fracture recognition | 3 months

SECONDARY OUTCOMES:
Secondary outcomes include BMD testing, diagnosis of osteoporosis, knowledge, and quality of life. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R. Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Kim N, Rowe BH, Raymond G, Jen H, Colman I, Jackson SA, Siminoski KG, Chahal AM, Folk D, Majumdar SR. Underreporting of vertebral fractures on routine chest radiography. AJR Am J Roentgenol. 2004 Feb;182(2):297-300. doi: 10.2214/ajr.182.2.1820297. PMID 14736649
- [Background] Majumdar SR, Kim N, Colman I, Chahal AM, Raymond G, Jen H, Siminoski KG, Hanley DA, Rowe BH. Incidental vertebral fractures discovered with chest radiography in the emergency department: prevalence, recognition, and osteoporosis management in a cohort of elderly patients. Arch Intern Med. 2005 Apr 25;165(8):905-9. doi: 10.1001/archinte.165.8.905. PMID 15851642
- [Result] Majumdar SR, McAlister FA, Johnson JA, Bellerose D, Siminoski K, Hanley DA, Qazi I, Lier DA, Lambert RG, Russell AS, Rowe BH. Interventions to increase osteoporosis treatment in patients with 'incidentally' detected vertebral fractures. Am J Med. 2012 Sep;125(9):929-36. doi: 10.1016/j.amjmed.2012.02.021. PMID 22938928
- [Result] Majumdar SR, Lier DA, McAlister FA, Rowe BH, Siminoski K, Hanley DA, Russell AS, Johnson JA. Cost-effectiveness of osteoporosis interventions for 'incidental' vertebral fractures. Am J Med. 2013 Feb;126(2):169.e9-17. doi: 10.1016/j.amjmed.2012.10.009. PMID 23331449